CLINICAL TRIAL: NCT00339391
Title: Socio-Environmental Determinants of Psychological Functioning, Mental Health and AIDS in Mali
Brief Title: Socioenvironmental Determinants of Psychological Functioning, Mental Health and AIDS in Mali
Status: Completed | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999901244; 01-M-N244
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2019-12-05 (Actual); Status verified 2016-11-30

CONDITIONS: AIDS; Stress
Keywords: Adjustment; Environmental Complexity; Mental Illness; Non-literate; West Africa; Stress; Knowledge; Mental Health; AIDS
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Mental Disorders; Psychological Well-Being

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other

SUMMARY:
This project is a collaboration between the Centre Regional de Medecine Traditionnelle (CRMT) of the Malian National Institute of Public Health Research (INRSP) and the Section on Socioenvironmental Studies (SSES). These units developed a three-pronged protocol reflecting their joint and individual concerns:

1. Effects of occupational complexity on psychological functioning. The project tests a theory derived from previous SSES research demonstrating that in industrialized societies doing relatively self-directed, substantively complex work increases self-directed orientations to self, society and family and promotes effective intellectual functioning. It uses sociological survey methodology to determine the generalizability of this theory to an essentially pre-literate, preindustrial society.
2. Effects of work-related stress on mental health. Earlier SSES work demonstrated that stressful work conditions lead to distress in industrialized societies. This project extends the investigation of these effects to a non-industrialized setting. It also extends the investigation of work-related stress to include work-related migration, resting a hypothesis that relates equally to SSES and CRMT concerns: that individuals from rural ethnic groups with a cultural tradition of work-related migration will show fewer mental health problems when migrating for nontraditional work than those from cultures without such a tradition. Mental health problems are assessed through: a) adaptations of standard survey-based psychological measures of components of distress, b) general and culture-specific survey-based psychiatric screening questions, and c) a psychiatric interview conducted by a CRMT psychiatrist trained in internationally accepted diagnostic procedures and knowledgeable about local cultures.
3. The effects of migration and cultural and socioeconomic factors on AIDS-related knowledge, attitudes and behaviors. The survey addresses concern regarding the degree of knowledge about the nature of AIDS among rural Malians who are relatively isolated from urban oriented sources of information about culturally non-traditional issues. It also examines how socio-cultural background and migration for work affect AIDS related attitudes and self-reported behaviors in an African society where estimates of HIV prevalence are still relatively low (less than 2%), compared to those of other sub-Saharan African countries.

Although these prongs are distinguishable, each requires a longitudinal design, a representative sample, extensive information about responders' social and cultural backgrounds, occupational histories, work conditions, and personal orientations and beliefs. Because of their overlapping theoretical approaches and methodological requirements, combining them in one project increases the richness and efficiency of the data collected for each.

DETAILED DESCRIPTION:
This project is a collaboration between the Centre Regional de Medecine Traditionnelle (CRMT) of the Malian National Institute of Public Health Research (INRSP) and the Section on Socioenvironmental Studies (SSES). These units developed a three-pronged protocol reflecting their joint and individual concerns:

1. Effects of occupational complexity on psychological functioning. The project tests a theory derived from previous SSES research demonstrating that in industrialized societies doing relatively self-directed, substantively complex work increases self-directed orientations to self, society and family and promotes effective intellectual functioning. It uses sociological survey methodology to determine the generalizability of this theory to an essentially pre-literate, preindustrial society.
2. Effects of work-related stress on mental health. Earlier SSES work demonstrated that stressful work conditions lead to distress in industrialized societies. This project extends the investigation of these effects to a non-industrialized setting. It also extends the investigation of work-related stress to include work-related migration, testing a hypothesis that relates equally to SSES and CRMT concerns: that individuals from rural ethnic groups with a cultural tradition of work-related migration will show fewer mental health problems when migrating for nontraditional work than those from cultures without such a tradition. Mental health problems are assessed through: a) adaptations of standard survey-based psychological measures of components of distress, b) general and culture-specific survey-based psychiatric screening questions, and c) a psychiatric interview conducted by a CRMT psychiatrist trained in internationally accepted diagnostic procedures and knowledgeable about local cultures.
3. The effects of migration and cultural and socioeconomic factors on AIDS-related knowledge, attitudes and behaviors. The survey addresses concern regarding the degree of knowledge about the nature of AIDS among rural Malians who are relatively isolated from urban oriented sources of information about culturally non-traditional issues. It also examines how socio-cultural background and migration for work affect AIDS related attitudes and self-reported behaviors in an African society where estimates of HIV prevalence are still relatively low (less than 2%), compared to those of other sub-Saharan African countries.

Although these prongs are distinguishable, each requires a longitudinal design, a representative sample, extensive information about responders' social and cultural backgrounds, occupational histories, work conditions, and personal orientations and beliefs. Because of their overlapping theoretical approaches and methodological requirements, combining them in one project increases the richness and efficiency of the data collected for each.

The division of responsibility between SSES and CRMT is as follows:

1. The survey questionnaire is the product of SSES/CRMT collaboration. It has been check by Malian linguists, extensively pretested by CRMT, and found feasible to administer and likely to provide highly reliable data with sufficient variance to permit the testing of our hypotheses. The project has been independently review and approved by the relevant Malian IRB the Ethics Committee and the Medical School of the University of Mali.
2. Data Collection involves conducting structured sociological interviews with representative rural samples from three Malian ethnic groups, carrying out psychiatric interviews with respondents who fail the psychiatric screen. The collection, processing and coding of the data is the responsibility of CRMT.
3. Data Analysis is primarily the responsibility of the SSES, which receives the data in a form in which individual respondents cannot be identified.

ELIGIBILITY:
* INCLUSION CRITERIA:

The study sample is a representative sample, based on Malian census data, of approximately 1000 respondents, age 16-50, drawn equally from each of the three generally pre-literate ethnic groups - the Dogon, the Peulh and the Bozo.

EXCLUSION CRITERIA:

Villages must not have heavily visited tourist attractions.

Ages: 16 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1002 (Actual)
Dates: Start 2001-08-19; Study Completion 2016-11-30

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Merikangas, Ph.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- Centre Regional de Medecine Traditionnelle, Bamako, Mali

REFERENCES:
- [Background] Kessler RC, Zhao S, Blazer DG, Swartz M. Prevalence, correlates, and course of minor depression and major depression in the National Comorbidity Survey. J Affect Disord. 1997 Aug;45(1-2):19-30. doi: 10.1016/s0165-0327(97)00056-6. PMID 9268772
- [Background] Maiga MY, Diarra B, Guindo A, Maiga YI, Fofano O, Bougoudogo F. [Seroprevalence of human immunodeficiency virus infection (HIV) in Mali on 3,496 sera]. Bull Soc Pathol Exot. 1993;86(1):16-20. French. PMID 8504258